CLINICAL TRIAL: NCT03582930
Title: Aerosolized Infasurf Treatment Protocol: Aerosolized Infasurf for Spontaneously Breathing Patients With Early RDS (AERO-03)
Status: No longer available | Type: Expanded Access
Sponsor: ONY (Industry)
Responsible Party: Sponsor
Other Study IDs: Aero-03
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-10

CONDITIONS: Neonatal Respiratory Distress
Keywords: Infasurf; Surfactant; RDS; Respiratory Distress Syndrome; Aerosolized; Nebulized; Inhaled; Pre-term; Premature
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Distress Syndrome; Respiratory Aspiration; Premature Birth

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Combination Product: Infasurf Aero — Aerosolization of Infasurf administered to premature babies suffering from RDS. Successful administration of Infasurf by aerosolization will provide two important benefits for patients. (1) endotracheal intubation may be able to be avoided in some patients, and (2) the adverse events at instillation due to filling the airway with liquid and interrupting breathing may be diminished or abolished.

SUMMARY:
Surfactant replacement therapy can be life-saving for newborn infants born with symptomatic lung surfactant deficiency causing Respiratory Distress Syndrome (RDS). Currently, such therapy requires instillation of a liquid suspension into the trachea through an endotracheal tube. Endotracheal intubations have undesirable adverse effects on fragile premature infants. Instilling surfactant as a liquid suspension into the lung is associated with adverse events due to interruption of breathing in patients who already have respiratory insufficiency. This treatment protocol is expanded access that offers the opportunity for patients to receive aerosolized Infasurf prior to FDA acting on ONY Biotech's application for approval for commercial marketing of aerosolized Infasurf.

DETAILED DESCRIPTION:
This Treatment Protocol will offer patients access to aerosolized Infasurf therapy at the time RDS is diagnosed if a patient is <12 hours of age and has not previously received liquid surfactant, or is <24 hours of age, and received liquid surfactant in the first hour after birth, was extubated and RDS is worsening. Parents must give informed consent. Up to 2 repeat doses of aerosolized Infasurf can be administered. Aerosolized Infasurf must be administered as described in the protocol. Adverse events at administration (if any) and all serious adverse events related or possibly related the aerosolized Infasurf therapy will be extracted from the medical record and reported to the sponsor, ONY Biotech. A copy of the discharge summary of patients will be collected by the sponsor using HIPAA compliant methodology for generation of a data set that will characterize adverse events and other efficacy and safety data.

ELIGIBILITY:
Inclusion Criteria:

Two cohorts with different entry criteria are included. In cohort 1 are patients with a diagnosis of early RDS who are not intubated and have not received a liquid surfactant instillation. In cohort 2 are patients who received liquid surfactant in the first hour of life, have been extubated and whose RDS is worsening.

Cohort 1 Inclusion Criteria

1. NICU patient, <12 hours of age.
2. Clinical diagnosis of RDS, with or without chest X-ray data.
3. Inspired oxygen ≤40% to maintain adequate oxygen saturation.
4. Not intubated
5. Requiring: (a) nasal continuous positive airway pressure (nCPAP), or (b) high flow nasal cannula (≥2L/kg/min) (HFNC), or (c) non-invasive ventilation.

Cohort 2 Inclusion Criteria

1. NICU patient, <24 hours of age who received liquid surfactant at ≤ 1 hour of age and was extubated.
2. Clinical diagnosis of RDS, with or without chest X-ray data.
3. Inspired oxygen ≤40% to maintain adequate oxygen saturation.
4. Not intubated
5. Requiring: (a) nasal continuous positive airway pressure (nCPAP), or (b) high flow nasal cannula (≥2L/kg/min) (HFNC), or (c) non-invasive ventilation.

Exclusion Criteria:

* 1) Requires >40% inspired oxygen to maintain acceptable oxygenation 2) Requires endotracheal intubation. 3) A co-existing medical condition that makes aerosol administration contraindicated in the judgment of the attending physician.

Max Age: 42 Weeks | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cummings, MD, Study Chair — Albany Medical College
Locations (5):
- United States (5):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Sisters of Charity Hospital, Buffalo, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Utah Valley Hospital, Provo, Utah